CLINICAL TRIAL: NCT04522700
Title: Reconstruction of Maxillary and Midfacial Defects Using Latissimus Dorsi Scapular Free Flaps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: hassan harby mohamed (Other)
Responsible Party: Sponsor-Investigator, hassan harby mohamed, principal investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: scapular free flaps
Record Dates: First submitted 2020-08-17; First posted 2020-08-21 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Maxillary Neoplasms
MeSH Terms: conditions — Maxillary Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: scapular free flap — use of scapular free flap to reconstruction post maxillectomy defect to provide bony support

SUMMARY:
Bony reconstruction of the midface with free tissue transfer is complex and challenging due to structural considerations such as the need for orbital support, patency of the nasal cavity, restoration of the palate and alveolus and skull base support when needed. As a result, bony reconstruction is important especially for patients who experience diplopia, hypoglobus and enophthalmos postoperatively.

Orocutaneous and nasocutaneous fistulae and infection due to communication with the oral cavity or sinuses are also common complication . Finally, cosmetic deformities from inadequate projection are also a concern.

Cosmetic and functional outcomes are improved with bony reconstruction as it is able to provide rigid support of key structures, restoration of contour, affords the possibility of dental rehabilitation and is less likely to contract significantly following radiation treatment.

Subscapular system free flaps (SF) are uniquely suited to address the needs of midface reconstruction. A substantial amount of bone can be harvested from the lateral scapular border and scapular tip, each with different shapes and thicknesses. Chimeric flaps can be harvested in various combinations, adding Para scapular and scapular skin paddles, latissimus muscle (with or without skin), serratus muscle and rib. Additionally, due to the vascular organization of this network, these components can be harvested off separate pedicles, offering great flexibility and freedom of movement relative to each other .

DETAILED DESCRIPTION:
reconstruction of defects post maxiilectomy by scapular free flaps

ELIGIBILITY:
Inclusion Criteria:

1. All patients post maxillectomy due to benign maxillary lesions.
2. All patients post maxillectomy with malignant maxillary swelling with no distant metastases.
3. All patients which implants are needed after surgery for head and neck neoplasia .

Exclusion Criteria:

1. Oropharyngeal, Nasopharyngeal, and Hypopharyngeal cancers, and lip cancers;.
2. Recurrent tumors resulting in implant loss.
3. Previous free flap harvest from scapula.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-25 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
reconstruction and restoration of facial contour. | 6 month
  reconstruction of the maxilla by provide rigid bony support post maxillectomy with measurement of graft taken and union occur by follow up with MSCT of the facial bone with 3D film .

CONTACTS AND LOCATIONS:
Overall Officials: hassan harby, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Sarukawa S, Kamochi H, Noguchi T, Sunaga A, Uda H, Mori Y, Nishino H, Yoshimura K. Free-flap surgical correction of facial deformity after anteromedial maxillectomy. J Craniomaxillofac Surg. 2017 Sep;45(9):1573-1577. doi: 10.1016/j.jcms.2017.06.020. Epub 2017 Jul 6. PMID 28747264